CLINICAL TRIAL: NCT04535037
Title: A Phase IV, Single-blind, Randomised, Controlled, Multi-country Study to Evaluate the Immunogenicity and Safety of GSK's Infanrix Hexa (DTPa-HBV-IPV/Hib) Versus MCM Vaccine BV's Vaxelis (DTaP5-HBV-IPV Hib), When Administered Intramuscularly According to a 2-, 4- and 12-month Schedule in Healthy Infants and Toddlers
Brief Title: A Study to Evaluate Immunogenicity and Safety of GlaxoSmithKline (GSK)'s Infanrix Hexa Vaccine (DTPa-HBV-IPV/Hib) Versus MCM Vaccine BV's Vaxelis Vaccine (DTaP5-HBV-IPV-Hib) in Healthy Infants and Toddlers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 212645; 2019-002988-10 (EudraCT Number)
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Diphtheria
Keywords: Primary immunization; Immunogenicity; Safety; Diphtheria; Tetanus; Acellular pertussis; Hepatitis B; Inactivated poliovirus; Haemophilus influenzae type b
MeSH Terms: conditions — Diphtheria; Tetanus; Hepatitis B; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Vaxelis; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infanrix Hexa (Experimental): All subjects in this group received 3 doses (2 primary doses and 1 booster dose) of DTPa-HBV-IPV/Hib vaccine co-administered with 3 doses of pneumococcal 13 valent conjugate vaccine at 2, 4, and 12 months of age.
  Interventions: Biological: DTPa-HBV-IPV/Hib; Biological: Pneumococcal 13-valent conjugate vaccine
- Vaxelis (Active Comparator): All subjects in this group received 3 doses (2 primary doses and 1 booster dose) of DTaP5 HBV IPV Hib vaccine co-administered with 3 doses of pneumococcal 13 valent conjugate vaccine at 2, 4, and 12 months of age.
  Interventions: Biological: DTaP5-HBV-IPV-Hib; Biological: Pneumococcal 13-valent conjugate vaccine

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib — 3 doses (1 each at 2, 4 and 12 months of age) of DTPa-HBV-IPV/Hib vaccine administered by intramuscular injection into the right thigh
  Other Names: Infanrix hexa
  Arms: Infanrix Hexa
Biological: DTaP5-HBV-IPV-Hib — 3 doses (1 each at 2, 4 and 12 months of age) of DTaP5-HBV-IPV-Hib vaccine administered by intramuscular injection into the right thigh
  Other Names: Vaxelis
  Arms: Vaxelis
Biological: Pneumococcal 13-valent conjugate vaccine — 3 doses (1 each at 2, 4 and 12 months of age) of pneumococcal 13-valent conjugate vaccine administered by intramuscular injection into the left thigh
  Other Names: Prevenar 13

SUMMARY:
The purpose of this study was to assess the safety and immunogenicity of GSK's combined diphtheria, tetanus, acellular pertussis, hepatitis B, inactivated poliovirus and Haemophilus influenzae type b conjugate vaccine (DTPa-HBV-IPV/Hib) versus MCM Vaccine BV's DTaP5-HBV-IPV-Hib vaccine administered to healthy infants and toddlers, between 6 and 12 weeks of age at the time of first vaccination, based on a 2-, 4-, and 12-months of age vaccination schedule.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) (LAR[s]) who, in the opinion of the investigator, could and would comply with the requirements of the protocol (e.g., return for follow-up visits).
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* A male or female child between and including 6 and 12 weeks of age (42 to 84 days) at the time of the first vaccination.
* Subject born after at least 37 weeks of gestation.
* Healthy subjects as established by the investigator based on medical history and the clinical examination before entering into the study.

Exclusion Criteria:

* Any clinical condition that, in the opinion of the investigator, might pose any risk to the subject due to participation in the study. As with other vaccines, administration of DTPa-HBV-IPV/Hib should be postponed in subjects suffering from acute severe febrile illness. The presence of a minor infection is not a contraindication.
* Known history of diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Hib diseases since birth.
* History of any reaction or hypersensitivity likely to be caused or exacerbated by any excipient or active component of the vaccine(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including malignancies, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects, as assessed by the investigator.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined via medical history including physical examination.
* Medical history of neurological disorder, including seizures.
* Previous vaccination for diphtheria, tetanus, pertussis, HBV, poliomyelitis, Hib diseases and previous vaccination against pneumococcal infection with pneumococcal conjugate vaccine, with the exception of a birth dose of HBV vaccine, which may have been given in accordance with local recommendations.
* Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study vaccine(s) during the period starting 30 days before the first dose of study vaccine(s) (Day -29 to Day 1), or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine(s) with the exception of administration of vaccines given as part of the national immunization schedule and as part of routine vaccination practice, e.g., rotavirus vaccine, that were allowed at any time during the study period. In case emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) would have been organized by public health authorities outside the routine immunization program, the time period described above could be reduced if necessary for that mass vaccination vaccine, provided this vaccine/product(s) is licensed and used according to its Product Information.
* Administration of long-acting immune-modifying drugs in the period starting 30 days before the first dose and at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives from birth or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine. For corticosteroids, this would mean prednisone ≥0.5 mg/kg/day (for paediatric subjects), or equivalent. Inhaled and topical steroids are allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or would have been exposed to an investigational or a non-investigational vaccine/product (drug or medical device).
* Child in care.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- Germany (10):
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Schönau am Königssee, Bavaria
  - GSK Investigational Site, Leipzig, Brandenburg
  - GSK Investigational Site, Wolfsburg, Lower Saxony
  - GSK Investigational Site, Hürth, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Bramsche
  - GSK Investigational Site, Erfurt
  - GSK Investigational Site, Mönchengladbach
- GSK Investigational Site, Milan, Italy
- Spain (8):
  - GSK Investigational Site, Málaga, Andalusia
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Boadilla Del Monte (Madrid)
  - GSK Investigational Site, Leganés
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Martinon-Torres F, Salamanca de la Cueva I, Horn M, Westerholt S, Bosis S, Meyer N, Cheuvart B, Virk N, Jakes RW, Duchenne M, Van den Steen P. Disparate kinetics in immune response of two different Haemophilus influenzae type b conjugate vaccines: Immunogenicity and safety observations from a randomized controlled phase IV study in healthy infants and toddlers using a 2+1 schedule. Hum Vaccin Immunother. 2024 Dec 31;20(1):2342630. doi: 10.1080/21645515.2024.2342630. Epub 2024 Apr 30. PMID 38687024

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infanrix Hexa | Vaxelis
Started | 249 | 251
Completed | 237 | 233
Not Completed | 12 | 18
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Migrated / moved from the study area | 1 | 4
Not completed — Other | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix Hexa | Vaxelis | Total
Number analyzed (Participants) | 249 | 251 | 500
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.6 (1.17) | 8.6 (1.24) | 8.6 (1.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 135 | 240
  Male | 144 | 116 | 260
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 2 | 3
  American Indian or Alaska Native | 1 | 2 | 3
  Asian - Central / South Asian Heritage | 0 | 1 | 1
  Asian - East Asian Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 0 | 1 | 1
  White - Arabic / North African Heritage | 5 | 4 | 9
  White - Caucasian / European Heritage | 236 | 235 | 471
  Other-Unspecified | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations at Month 11, Based on Per Protocol Set (PPS)
Description: Anti-PRP antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in microgram per milliliter (μg/mL), as assessed by Enzyme-linked immunosorbent assay (ELISA).
Time Frame: At Month 11 (i.e., 1-month post-booster vaccination)
Population: The analysis was performed on the Per Protocol Set (PPS), which included all eligible subjects who received diphtheria, tetanus and acellular pertussis (DTPa)-combination study vaccines as per protocol, who had anti-PRP results post-vaccination, who complied with vaccination/blood draw intervals, without intercurrent conditions and without prohibited concomitant medication/vaccination and for whom immunogenicity data were available for specific timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 211 | 218
μg/mL | 11.61 [NA to NA] — As specified in the Statistical Analysis Plan, for the co-primary objectives, only geometric mean was calculated for anti-PRP antibody concentration and was adjusted for DTPa vaccination of the mother. | 12.66 [NA to NA] — As specified in the Statistical Analysis Plan, for the co-primary objectives, only geometric mean was calculated for anti-PRP antibody concentration and was adjusted for DTPa vaccination of the mother.
Statistical Analysis 1: Comparison: Infanrix Hexa vs Vaxelis; To demonstrate that the Haemophilus influenzae type b(Hib) response of Infanrix Hexa Group is non-inferior to the Vaxelis Group in terms of anti-PRP GMCs, 1 month post-booster vaccination; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit (LL) of the 2-sided 95% confidence interval (CI) of group GMC ratio (Infanrix Hexa over Vaxelis group) was above 0.5; The 95% CI for GMC ratio derived from an ANOVA model on log10 transformed concentration was used. GMC was adjusted for DTPA vaccination of the mother; Adjusted GMC Ratio = 0.917, 95% CI 2-sided [0.710 to 1.185]

2. Primary Outcome: Percentage of Subjects With Anti-PRP Antibody Concentrations Equal to or Above (≥) 5 µg/mL at Month 11, Based on PPS
Description: The percentage of subjects with anti-PRP antibody concentrations ≥5 µg/mL was reported, as assessed by ELISA.
Time Frame: At Month 11 (i.e., 1-month post-booster vaccination)
Population: The analysis was performed on PPS, which included all eligible subjects who received all DTPa-combination study vaccines as per protocol, who had anti-PRP results post-vaccination, who complied with vaccination/blood draw intervals, without intercurrent conditions and without prohibited concomitant medication/vaccination and for whom immunogenicity data were available for specific timepoints.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 211 | 218
Percentage of Participants | 75.4 | 81.7
Statistical Analysis 1: Comparison: Infanrix Hexa vs Vaxelis; To demonstrate that the Hib response in Infanrix Hexa group is non-inferior to Vaxelis Group in terms of percentage of subjects with anti-PRP antibody concentrations ≥ 5 µg/mL, 1 month post-booster vaccination; Test type: Non-Inferiority — Non-inferiority was demonstrated if the non inferiority of anti-PRP GMC ratio was met and the LL of the 2 sided 95% CI on group difference in the percentage (Infanrix Hexa over Vaxelis group) was more than -10%; The 2 sided 95% CI of group difference in seroconversion rate (Inv_group minus Com_group) was computed based on Miettinen and Nurminen method; Difference in Percentage = -6.30, 95% CI 2-sided [-14.10 to 1.49]

3. Primary Outcome: Anti-PRP Antibody Concentrations at Month 11, Based on the Exposed Set (ES)
Description: Anti-PRP antibody concentrations were presented as GMCs and expressed in μg/mL, as assessed by ELISA.
Time Frame: At Month 11 (i.e., 1-month post-booster vaccination)
Population: The analysis was performed on the Exposed Set (ES), which included all vaccinated subjects who were analysed according to the intervention they received at Dose 1 and for whom immunogenicity data were available for specific timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 175 | 228
μg/mL | 11.26 [NA to NA] — As specified in the Statistical Analysis Plan, for the co-primary objectives, only geometric mean was calculated for anti-PRP antibody concentration and was adjusted for DTPa vaccination of the mother. | 12.85 [NA to NA] — As specified in the Statistical Analysis Plan, for the co-primary objectives, only geometric mean was calculated for anti-PRP antibody concentration and was adjusted for DTPa vaccination of the mother.

4. Primary Outcome: Percentage of Subjects With Anti-PRP Antibody Concentrations ≥ 5 µg/mL at Month 11, Based on ES
Description: The percentage of subjects with anti-PRP antibody concentrations ≥5 µg/mL was reported, as assessed by ELISA.
Time Frame: At Month 11 (i.e., 1-month post-booster vaccination)
Population: The analysis was performed on the ES, which included all vaccinated subjects who were analysed according to the intervention they received at Dose 1 and for whom immunogenicity data were available for specific timepoints.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 175 | 186
Percentage of Participants | 75.4 | 81.6

5. Secondary Outcome: Percentage of Subjects With Anti-PRP Antibody Concentration ≥ 0.15 µg/mL
Description: The percentage of subjects with anti-PRP antibody concentration equal to or above the threshold for short-term protection was reported. The threshold for short-term protection is 0.15 µg/mL.
Time Frame: At Month 3 (i.e., 1-month post-primary vaccination), Month 10 (i.e., pre-booster) and Month 11 (i.e., 1-month post-booster vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 213 | 230
Percentage of Participants
  At month 3 | 79.8 [73.79 to 84.99] | 100 [98.41 to 100]
  At Month 10: number analyzed (Participants) | 206 | 216
  At Month 10 | 61.2 [54.14 to 67.86] | 94.4 [90.50 to 97.10]
  At Month 11: number analyzed (Participants) | 211 | 218
  At Month 11 | 99.5 [97.39 to 99.99] | 99.5 [97.47 to 99.99]

6. Secondary Outcome: Percentage of Subjects With Anti-PRP Antibody Concentrations ≥ 1.0 µg/mL
Description: The percentage of subjects with anti-PRP antibody concentration equal to or above the threshold for long-term protection was reported. The threshold for long-term protection is 1.0 µg/mL.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 213 | 230
Percentage of Participants
  At Month 3 | 30.5 [24.41 to 37.18] | 92.2 [87.91 to 95.30]
  At Month 10: number analyzed (Participants) | 206 | 216
  At Month 10 | 13.1 [8.82 to 18.49] | 69.0 [62.35 to 75.08]
  At Month 11: number analyzed (Participants) | 211 | 218
  At Month 11 | 97.2 [93.91 to 98.95] | 94.5 [90.58 to 97.12]

7. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Anti-PRP antibody concentrations were presented as GMCs and expressed in μg/mL, as assessed by ELISA.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 213 | 230
μg/mL
  At Month 3 | 0.5 [0.41 to 0.62] | 11.3 [9.35 to 13.60]
  At Month 10: number analyzed (Participants) | 206 | 216
  At Month 10 | 0.2 [0.19 to 0.28] | 1.9 [1.56 to 2.26]
  At Month 11: number analyzed (Participants) | 211 | 218
  At Month 11 | 12.0 [9.96 to 14.34] | 12.9 [10.75 to 15.55]

8. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: AEs are defined as any untoward medical occurrence in a subject or subjects, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: During the 31-day (Days 1-31) follow-up period after each vaccination (vaccines administered at 2,4 and 12 months of age)
Population: The analysis was performed on the ES, which included all vaccinated subjects who were analysed according to the intervention they received at Dose 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 249 | 251
Participants | 178 | 199

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: A SAEs is defined as any untoward medical occurrence that, at any dose, result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect.
Time Frame: Throughout the entire period of the study (from Day 1 up to study end [Month 11])
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa | Vaxelis
Number analyzed (Participants) | 249 | 251
Participants | 14 | 10

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected throughout the entire period of the study (from Day 1 up to study end [Month 11]). Non Serious AEs (Other AEs) were collected during the 31 days follow-up period after each vaccination (vaccines administered at 2,4 and 12 months of age).
Arm/Group | Infanrix Hexa | Vaxelis
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/251
Serious Adverse Events (participants affected / at risk) | 14/249 | 10/251
Other Adverse Events (participants affected / at risk) | 178/249 | 199/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix Hexa (N=249) | Vaxelis (N=251)
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Abscess neck (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 2 | 3
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 2
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 3
Rhinovirus infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Enterovirus test positive (Investigations) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 2 | 0
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infanrix Hexa (N=249) | Vaxelis (N=251)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Microcephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Plagiocephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Astigmatism (Eye disorders) | 1 (1) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 3 (3) | 1 (1)
Eye haematoma (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Hypermetropia (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 9 (10)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 15 (20) | 16 (19)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 4 (4)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 3 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 8 (10) | 5 (5)
Administration site haemorrhage (General disorders) | 0 (0) | 1 (1)
Administration site pain (General disorders) | 0 (0) | 1 (1)
Crying (General disorders) | 5 (5) | 7 (7)
Discomfort (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 2 (2) | 3 (4)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1)
Induration (General disorders) | 1 (1) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Injection site discomfort (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 6 (8) | 8 (9)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 3 (3) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 6 (7) | 8 (8)
Injection site swelling (General disorders) | 7 (8) | 8 (11)
Injection site warmth (General disorders) | 0 (0) | 2 (2)
Irritability postvaccinal (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 2 (3) | 3 (3)
Nodule (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (3)
Peripheral swelling (General disorders) | 4 (4) | 4 (4)
Pyrexia (General disorders) | 103 (181) | 132 (237)
Swelling (General disorders) | 1 (1) | 1 (1)
Vaccination site erythema (General disorders) | 0 | 2
Vaccination site granuloma (General disorders) | 0 (0) | 1 (2)
Vaccination site induration (General disorders) | 0 (0) | 2 (2)
Vaccination site swelling (General disorders) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 3 (3)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 4 (4) | 3 (3)
Bronchitis (Infections and infestations) | 6 (7) | 5 (5)
Candida nappy rash (Infections and infestations) | 2 (2) | 2 (2)
Conjunctivitis (Infections and infestations) | 14 (14) | 14 (15)
COVID-19 (Infections and infestations) | 14 (14) | 9 (9)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 2 (2) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 9 (9) | 10 (11)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 2 (2)
Herpangina (Infections and infestations) | 1 (1) | 2 (2)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 5 (5) | 4 (4)
Nasopharyngitis (Infections and infestations) | 6 (7) | 14 (14)
Oral candidiasis (Infections and infestations) | 4 (4) | 5 (5)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 5 (5) | 6 (6)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal disease (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 6 (8)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 3 (3)
Rhinitis (Infections and infestations) | 2 (2) | 5 (5)
Roseola (Infections and infestations) | 1 (1) | 0 (0)
Subglottic laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 18 (22) | 20 (24)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 4 (4)
Viral rash (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 5 (6) | 6 (6)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electric shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hair-thread tourniquet syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 1 (1) | 2 (2)
Body temperature decreased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 3 (3) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 5 (5)
Hypoferritinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Head titubation (Nervous system disorders) | 0 (0) | 1 (1)
Hypertonia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 5 (5)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 31 (48) | 37 (56)
Restlessness (Psychiatric disorders) | 8 (14) | 13 (18)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Genital labial adhesions (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 6 (7) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT04535037/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT04535037/SAP_001.pdf